CLINICAL TRIAL: NCT07206108
Title: A Multicenter, Randomized Controlled, Single-blind, Non-inferiority Clinical Trial of Modified Endocrown and Personalized Post Core Combined With Full Crown for Large-area Tooth Defects After Root Canal Treatment
Brief Title: Clinical Trial of Modified Endocrown and Personalized Post-core and Crown for Large-area Tooth Defects After Root Canal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Stomatological Hospital of Southern Medical University (Unknown); Guanghua Stomatological Hospital, Sun Yat-sen University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2025-270
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Root Canal Infection; Tooth Defect; Post and Core Technique
Keywords: Modified endocrown; endocrown; personalized post and core combined with full crown; CAD/CAM; Teeth defect; Restoration of large-area defective teeth after root canal treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified endocrown (Experimental): 1. preparation of residual crown: A. occlusal surface reduction of about 1.5-2mm, hole edge angle rounded;B. root canal orifice extension: remove all decay, remove root canal filling material 2mm below the root canal orifice;C. pulp cavity wall formation: form 2-5° extension of the wall, if there is a concave with mobile resin restoration.
  2. model design: use CEREC digital intraoral scanner
  3. Cutting: using CEREC MCX CAD/CAM system, cutting lithium disilicate glass ceramic block (IPSe. max CAD), fitting modified pulp cavity retention crown on teeth, adjusting occlusion, post-treatment of restoration, bonding with all-acid etching resin cement.
  Interventions: Procedure: modified endocrown
- Personalized pile core combined with full crown (No Intervention): 1. Coronal preparation: Remove all existing restorations and carious tissue, eliminate unsupported enamel, flatten the root surface, establish the definitive margin, and ensure the dentin ferrule is ≥1 mm thick and ≥1.5 mm high.
  2. Post-space preparation: Set post depth at ⅔-¾ of root length (≥ clinical crown length) using the working-length and periapical radiograph; remove obturation material to this depth with a pilot drill, leaving ≥4 mm apical seal.
  3. Core restoration: Take a polyether impression of the post space, have a Co-Cr post-and-core fabricated, lute it with self-adhesive resin cement (RelyX U100/U200; 3M-ESPE), then prepare the core for a full crown.
  4. Full-crown fabrication: Record a polyether impression/optical scan, have a lithium-disilicate ceramic crown (IPS e.max CAD) milled, try-in and adjust, then cement definitively with the same self-adhesive resin cement following manufacturer instructions.

INTERVENTIONS:
Procedure: modified endocrown — Combining the advantages of post-core crown and endocrown, an modified endocrown was designed
  Arms: modified endocrown

SUMMARY:
This study intends to adopt a multicenter, randomized controlled, single-blind, non-inferiority clinical trial design. 246 premolars that meet the inclusion criteria after complete root canal treatment will be selected from the clinical practice and randomly divided into two groups. One group will be restored with the modified endocrown, and the other group will be restored with personalized post and core combined with full crown. Follow-up visits were conducted at 6 months, 1 year and 2 years after the operation respectively. Through clinical and imaging examinations, the survival rates of the two different restorations were evaluated and used as the main evaluation indicators to fill the gap in efficacy data of the modified endocrown in clinical applications, providing a strong evidence-based medical basis for subsequent restoration improvement and standardized application.

ELIGIBILITY:
Inclusion Criteria:

* 1: The affected tooth was a premolar that had undergone complete root canal treatment for two weeks. Both imaging and clinical examinations indicated no abnormal periapical reactions.

  2: The oral hygiene condition is good. There is no periodontitis or combined periodontal and endodontic lesions with a probing depth greater than 4mm. There are no severe oral bad habits (such as smoking more than 20 cigarettes per day, chewing betel nuts, etc.)

  3: At least 50% of the crown structure should be retained, or at least two crown walls should be retained, and the tooth defect should not be located under the gums or can be aligned with the gums or located above the gums through crown lengthening surgery.

  4: The affected tooth has sufficient root length to ensure a pedicle-crown ratio of at least 1:1 and a root tip closure of at least 3 mm.

  5: The occlusal function is normal.

  6: Treated premolars will not be used as abutments for FPD or RPD restoration.

Exclusion Criteria:

* 1: Root canal retreatment of the affected tooth.

  2: Loosening > I °, alveolar bone resorption exceeds 1/3 of the root length.

  3: Loss of adjacent teeth and occlusal teeth.

  4: The patient is in the preconception period and the pregnancy period.

  5: Patients with night bruxism, deep overbite, tight occlusion or severe limited mouth opening, and temporomandibular joint diseases.

  6: Patients who have a history of chemotherapy or radiotherapy in the head and neck region within 5 years, suffer from severe systemic and organic diseases, have physical disabilities or mental illnesses that affect oral hygiene care, or have received drug treatment that may affect or promote bone metabolism within the past 3 months.

  7: The affected tooth has imaging manifestations of absorption inside and outside the root, or the anatomical morphology of the root and root canal is poor, such as short and small roots, curved root canals, small roots or residual roots that cannot meet the cord-to-root ratio standard for pile-core crown restoration.

  8: The researchers consider other situations that are not suitable for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
survival rate | 6 month、1 year、2 years
  To evaluate secondary caries, proximal anatomy, gingival health, tooth integrity, marginal adaptability, fracture and retention, and radiographic results of the restoration, and to calculate FDI scores for the above indicators according to the World Dental Federation evaluation criteria (FDI), calculate the survival rate of the restoration

SECONDARY OUTCOMES:
Tooth reserve volume | immediately
  After root canal treatment and before tooth preparation, each tooth was scanned by CEREC extraoral scanner before tooth preparation. Each tooth was scanned by CEREC extraoral scanner to obtain an original STL file A before tooth preparation. After tooth preparation, the original STL file A1 after tooth preparation was obtained. The files A and A1 were imported into reverse engineering software (GeomagicControlX2020; Geomagic Inc.), calculated and recorded the amount of tooth preparation tissue of each tooth, and finally statistically analyzed the amount of tooth preparation tissue of the two groups.
patient satisfaction | 2 years
  visual analogue scale，VAS
Adjust the amount of grinding tissue and the time of occlusal adjustment | immediately
  After the prostheses are made, the prostheses are scanned by CEREC extraoral scanner, and each prosthesis will obtain an original STL file B, which will be bonded and fixed, adjusted, and scanned again by the same scanner to obtain the final STL file B1 of the prosthesis. The files B and B1 will be imported into reverse engineering software (Geomagic Control X2020; Geomagic Inc., calculated the adjustment tissue volume of the restoration, recorded the adjustment time during the operation, and finally analyzed the adjustment tissue volume and adjustment time of the two groups of restoration statistically.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern Medical University, China, China

IPD SHARING:
Plan to Share IPD: No